CLINICAL TRIAL: NCT05047770
Title: A Phase III, Randomized, Open-label, Controlled, Multicenter Study to Evaluate the Immune Response and Safety of Both Herpes Zoster Subunit Vaccine in Healthy Adults Aged 50 Years and Older AND the Influenza Virus Vaccine in Healthy Adults Aged 18 Years and Older When Administered Sequentially or Coadministered With mRNA-1273 Booster Vaccination
Brief Title: A Study on the Immune Response and Safety of the Shingles Vaccine and the Influenza Vaccine When Either is Given to Healthy Adults at the Same Time or Following a COVID-19 Booster Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217670
Record Dates: First submitted 2021-09-15; First posted 2021-09-17 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Herpes Zoster
Keywords: COVID-19; Shingles; Influenza; Booster vaccination; HZ/su vaccine; Recombinant Zoster vaccine; Flu D-QIV vaccine; mRNA-1273 vaccine; Safety; Immunogenicity
MeSH Terms: conditions — Herpes Zoster; COVID-19; Influenza, Human | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Masking Description: Open-label study; participants randomly assigned to either the co-administration or sequential study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- HZ/suSeq Group (Active Comparator): Participants randomized to HZ/suSeq Group received one mRNA-1273 booster dose administered at Day 1, followed by the first dose of HZ/su vaccine administered at Week 2 and the second dose of HZ/su vaccine administered at Week 10.
  Interventions: Biological: HZ/su; Biological: mRNA-1273
- HZ/suCoAd Group (Experimental): Participants randomized to HZ/suCoAd Group received one mRNA-1273 booster dose co-administered with the first dose of HZ/su vaccine at Day 1, followed by the second dose of HZ/su vaccine administered at Week 8.
  Interventions: Biological: HZ/su; Biological: mRNA-1273
- FluD-QIVSeq Group (Active Comparator): Participants randomized to FluD-QIVSeq Group received one mRNA-1273 booster dose at Day 1, followed by one dose of Flu D-QIV vaccine at Week 2.
  Interventions: Combination Product: Flu D-QIV; Biological: mRNA-1273
- FluD-QIVCoAd Group (Experimental): Participants randomized to FluD-QIVCoAd Group received one mRNA-1273 booster dose co-administered with one dose of Flu D-QIV vaccine at Day 1.
  Interventions: Combination Product: Flu D-QIV; Biological: mRNA-1273

INTERVENTIONS:
Biological: HZ/su — 2 doses of HZ/su vaccine administered intramuscularly, either sequentially (HZ/suSeq Group) or simultaneously (HZ/suCoAd Group) with the mRNA-1273 booster dose. The second dose of HZ/su was administered 8 weeks after the first dose of HZ/su vaccine.
  Arms: HZ/suCoAd Group; HZ/suSeq Group
Combination Product: Flu D-QIV — 1 dose of Flu D-QIV vaccine administered intramuscularly, either sequentially (FluD-QIVSeq Group) or simultaneously (FluD-QIVCoAd Group) with the mRNA-1273 booster dose.
  Other Names: Flu Quadrivalent Influenza Vaccine
  Arms: FluD-QIVCoAd Group; FluD-QIVSeq Group
Biological: mRNA-1273 — 1 booster dose of mRNA-1273 vaccine administered intramuscularly at Day 1 (all groups).

SUMMARY:
The aim of this study was to evaluate the immune response and safety of both GlaxoSmithKline Biologicals SA's (GSK's) herpes zoster (HZ) subunit (su) vaccine in healthy adults 50 years of age (YOA) and older and quadrivalent seasonal influenza (Flu D-QIV) vaccine in healthy adults 18 YOA and older, when administered sequentially or co-administered with Moderna's mRNA-1273 booster vaccination against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Participants who in the opinion of the investigator, can and who will comply with the requirements of the protocol (e.g., completion of the eDiaries, return for follow-up visits).
* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* Age at study entry:

  * For HZ/su and mRNA-1273 booster cohort: A male or female aged 50 years or older at the time of randomization.
  * For Flu D-QIV and mRNA-1273 booster cohort: A male or female aged 18 years or older at the time of enrollment.
* Healthy participants or medically stable patients as established by medical history and clinical examination at screening. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrolment.
* Participants who have a documented previous mRNA-1273 primary vaccination series completed (i.e., both doses) at least 6 months prior to first vaccination.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, documented total hysterectomy, bilateral ovariectomy, or bilateral salpingectomy, or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * Has practiced effective contraception for 1 month prior to study intervention administration, and
  * Has a negative pregnancy test on the day of study intervention administration, and
  * Has agreed to continue effective contraception during the study until 2 months after completion of the study vaccination series.

Exclusion Criteria:

Medical conditions

* Any clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study or might confound post-study intervention administration safety assessments (e.g., tattoos overlying either study intervention administration site).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions, including a known history of severe allergic reaction (e.g., anaphylaxis) to any component of any of the study vaccines.
* Any history of Guillain-Barré syndrome.
* Any history of myocarditis or pericarditis.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history or physical examination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Hypersensitivity to latex.
* For HZ/su and mRNA-1273 booster cohort: history of Herpes Zoster.

Prior/concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study intervention(s) during the period beginning 30 days before the first dose of study intervention(s) (Day -29 to Day 1), or their planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before first dose and ending 30 days after the last dose of study intervention administration. However, for HZ/su and mRNA-1273 booster cohort: licensed pneumococcal vaccines and non-replicating vaccines (i.e., inactivated and subunit vaccines, including inactivated and subunit influenza vaccines, with or without adjuvant for seasonal or pandemic flu) may be administered up until 8 days prior to dose 1 of HZ/su and/or dose 2 of HZ/su and/or at least 14 days after any dose of HZ/su. For Flu D-QIV and mRNA-1273 booster cohort: licensed pneumococcal vaccines and non-replicating vaccines (i.e., inactivated and subunit vaccines, other than influenza vaccines) may be administered up until 8 days prior to dose 1 of Flu D-QIV and/or at least 30 days after any dose of Flu D-QIV. For time interval between other routine vaccines with mRNA-1273 booster dose (administered in the study), local guidelines must be followed.

In case emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is organized by public health authorities outside the routine immunization program, the time period described above can be reduced if necessary for that mass vaccination vaccine, provided this vaccine is licensed and used according to its Product Information.

* Administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first dose of study intervention(s) up to 1 month post last dose or planned administration during the study period.
* Prior planned or chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine. For corticosteroids, this will mean more than 14 days in total of prednisone ≥20 mg/day or equivalent is not allowed. Inhaled, intra-articular and topical steroids are allowed.
* For HZ/su and mRNA-1273 booster cohort: Previous vaccination against Herpes Zoster with the exception of receipt of live attenuated HZ vaccine.
* For Flu D-QIV and mRNA-1273 booster cohort: Administration of a seasonal influenza vaccine during the 6 months preceding entry into the study.
* Prior administration of an investigational or licensed coronavirus (SARS-CoV, MERS-CoV, SARS-CoV-2) vaccine except for mRNA-1273 vaccine.
* Any contraindication to the study intervention(s).

Prior/concurrent clinical study experience

• Planning to or concurrently participating in another clinical study (including current / planned simultaneous participation in another interventional study to prevent or treat COVID-19), at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine / product (drug or medical device).

Other exclusions

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 2 months following last study vaccination.
* Indications of drug abuse or excess alcohol use as deemed by investigator to potentially confound safety assessments or render participant unable or unlikely to adhere to protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2013 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (43):
- United States (43):
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Atlantis, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, El Dorado, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Biloxi, Mississippi
  - GSK Investigational Site, Fremont, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Norman, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Yukon, Oklahoma
  - GSK Investigational Site, Grants Pass, Oregon
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Cedar Park, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Cheney, Washington
  - GSK Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Derived] Naficy A, Kuxhausen A, Seifert H, Hastie A, Leav B, Miller J, Anteyi K, Mwakingwe-Omari A. No immunological interference or concerns about safety when seasonal quadrivalent influenza vaccine is co-administered with a COVID-19 mRNA-1273 booster vaccine in adults: A randomized trial. Hum Vaccin Immunother. 2024 Dec 31;20(1):2327736. doi: 10.1080/21645515.2024.2327736. Epub 2024 Mar 21. PMID 38513689
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954
- [Derived] Naficy A, Kuxhausen A, Pirrotta P, Leav B, Miller J, Anteyi K, Danier J, Breuer T, Mwakingwe-Omari A. No Immunological Interference or Safety Concerns When Adjuvanted Recombinant Zoster Vaccine Is Coadministered With a Coronavirus Disease 2019 mRNA-1273 Booster Vaccine in Adults Aged 50 Years and Older: A Randomized Trial. Clin Infect Dis. 2023 Nov 11;77(9):1238-1246. doi: 10.1093/cid/ciad361. PMID 37335963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 47 centers in the United States.
Pre-assignment Details: Out of 2013 participants enrolled in the study, 468 were screen failures and 1545 were randomized to study groups. Out of 1545 randomized participants, only 1534 received at least 1 dose of study vaccine, were included in the Exposed Set and started the study.
Period: Overall Study
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Started | 272 | 267 | 497 | 498
Completed | 249 | 252 | 478 | 473
Not Completed | 23 | 15 | 19 | 25
Not completed — Withdrawal by Subject | 15 | 10 | 6 | 12
Not completed — Lost to Follow-up | 7 | 5 | 12 | 13
Not completed — Other | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group | FluD-QIVSeq Group | FluD-QIVCoAd Group | Total
Number analyzed (Participants) | 272 | 267 | 497 | 498 | 1534
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (8.38) | 62.5 (8.77) | 48.7 (16.10) | 49.5 (15.45) | 55.7 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 155 | 302 | 274 | 880
  Male | 123 | 112 | 195 | 224 | 654
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 1 | 4 | 5 | 10
  ASIAN | 2 | 1 | 17 | 15 | 35
  BLACK OR AFRICAN AMERICAN | 13 | 12 | 28 | 30 | 83
  WHITE | 247 | 250 | 436 | 435 | 1368
  MIXED ORIGIN | 4 | 1 | 5 | 4 | 14
  OTHER, UNSPECIFIED | 6 | 2 | 7 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Anti-glycoprotein E (gE) Antibody Concentrations Expressed as Geometric Mean Concentrations (GMCs) in HZ/suSeq and HZ/suCoAd Groups, and Between-group Ratios
Description: Anti-gE antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as GMCs in milli-international units per milliliter (mIU/mL).
Time Frame: At 1 month post-dose 2 of HZ/su vaccine administration (Week 14 for HZ/suSeq group and Week 12 for HZ/suCoAd group)
Population: HZ/su Per Protocol Set included all participants who met all eligibility criteria, received all doses as per assignment, for whom administration site of study vaccine was known, who did not receive any other prohibited concomitant intervention, did not meet any of the criteria for elimination up to blood sample collection post-HZ/su Dose 2, and with immunogenicity data available for the specified analysis at the specified time point post-HZ/su Dose 2.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 228 | 230
mIU/mL | 47434.82 [43306.87 to 51956.24] | 47599.82 [43960.57 to 51540.33]
Statistical Analysis 1: Comparison: HZ/suSeq Group vs HZ/suCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 2 doses of HZ/su vaccine when the first dose of HZ/su vaccine was co-administered with the mRNA-1273 booster dose compared to HZ/su vaccine administered alone, in terms of anti-gE GMCs, at 1 month post-dose 2 of HZ/su vaccine administration (Week 14 for HZ/suSeq group and Week 12 for HZ/suCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the upper limit (UL) of the 95% confidence interval (CI) of the adjusted GMC ratio between HZ/suSeq group and HZ/suCoAd group for anti-gE antibody concentration was below (<) 1.5; ANCOVA; GMC Ratio = 1.01, 95% CI 2-sided [0.89 to 1.13]

2. Primary Outcome: Anti-S Protein Antibody Concentrations Expressed as GMCs in HZ/suSeq and HZ/suCoAd Groups, and Between-group Ratios
Description: Anti-S antibody concentrations were determined by Multiplex Electrochemiluminescence assay and expressed as GMCs in arbitrary units per milliliter (AU/mL).
Time Frame: At 1 month post-mRNA-1273 booster dose administration (Week 4 for both HZ/suSeq and HZ/suCoAd groups)
Population: mRNA-1273 Per Protocol Set (for HZ/su groups) included all participants who met all eligibility criteria, received all doses as per assignment, for whom administration site of study vaccine was known, who did not receive any other prohibited concomitant intervention, did not meet any of the criteria for elimination up to blood sample collection post-mRNA-1273 dose, and with immunogenicity data available for the specified analysis at the specified time point post-mRNA-1273 dose.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 247 | 247
AU/mL | 618638.92 [526014.86 to 727572.81] | 567728.74 [513530.08 to 627647.61]
Statistical Analysis 1: Comparison: HZ/suSeq Group vs HZ/suCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of mRNA-1273 booster when the first dose of HZ/su vaccine was co-administered with the mRNA-1273 booster dose compared to mRNA-1273 booster dose administered alone, in terms of anti-S protein GMCs, at 1 month post-mRNA-1273 booster dose administration (at Week 4 for both HZ/suSeq and HZ/suCoAd groups); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the adjusted GMC ratio between HZ/suSeq group and HZ/suCoAd group for anti-S protein antibody concentration was <1.5; ANCOVA; GMC Ratio = 1.09, 95% CI 2-sided [0.90 to 1.32]

3. Primary Outcome: Anti-hemagglutinin Inhibition (HI) Antibody Titers Expressed as Geometric Mean Titers (GMTs) Against the 4 Influenza Strains in Flu D-QIV Vaccine in FluD-QIVSeq and FluD-QIVCoAd Groups, and Between-group Ratios
Description: Antibody titers against the 4 influenza strains (A/H1N1 strain, A/H3N2 strain, B/Victoria lineage and B/Yamagata lineage) included in the FLU D-QIV vaccine were determined by hemagglutination inhibition and expressed as GMTs.
Time Frame: At 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group)
Population: Flu D-QIV Per Protocol Set included all participants who met all eligibility criteria, received all doses as per assignment, for whom administration site of study vaccine was known, who did not receive any other prohibited concomitant intervention, did not meet any of the criteria for elimination during the study through the last blood sample for the group, and with immunogenicity data available for the specified analysis at the specified time point post-Flu D-QIV dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 454 | 462
Titers
  A/H1N1: number analyzed (Participants) | 453 | 461
  A/H1N1 | 598.62 [535.51 to 669.17] | 577.77 [517.80 to 644.68]
  A/H3N2 | 268.32 [242.17 to 297.30] | 280.26 [252.47 to 311.11]
  B/Victoria lineage | 48.00 [43.19 to 53.34] | 47.21 [42.47 to 52.49]
  B/Yamagata lineage | 55.30 [49.64 to 61.61] | 48.74 [43.83 to 54.21]
Statistical Analysis 1: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of Flu D-QIV vaccine when co-administered with mRNA-1273 booster dose compared to Flu D-QIV vaccine administered alone, in terms of anti-HI GMTs against the A/H1N1 influenza strain included in the Flu D-QIV vaccine, at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the adjusted GMT ratio between FluD-QIVSeq group and FluD-QIVCoAd group for anti-HI antibody titer was <1.5 for the A/H1N1 influenza strain; ANCOVA; GMT Ratio = 1.02, 95% CI 2-sided [0.89 to 1.18]
Statistical Analysis 2: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of Flu D-QIV vaccine when co-administered with mRNA-1273 booster dose compared to Flu D-QIV vaccine administered alone, in terms of anti-HI GMTs against the A/H3N2 influenza strain included in the Flu D-QIV vaccine, at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the adjusted GMT ratio between FluD-QIVSeq group and FluD-QIVCoAd group for anti-HI antibody titer was <1.5 for the A/H3N2 influenza strain; ANCOVA; GMT Ratio = 0.93, 95% CI 2-sided [0.82 to 1.05]
Statistical Analysis 3: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of Flu D-QIV vaccine when co-administered with mRNA-1273 booster dose compared to Flu D-QIV vaccine administered alone, in terms of anti-HI GMTs against the B/Victoria lineage influenza strain included in the Flu D-QIV vaccine, at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the adjusted GMT ratio between FluD-QIVSeq group and FluD-QIVCoAd group for anti-HI antibody titer was <1.5 for the B/Victoria lineage influenza strain; ANCOVA; GMT Ratio = 1.00, 95% CI 2-sided [0.89 to 1.14]
Statistical Analysis 4: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of Flu D-QIV vaccine when co-administered with mRNA-1273 booster dose compared to Flu D-QIV vaccine administered alone, in terms of anti-HI GMTs against the B/Yamagata lineage influenza strain included in the Flu D-QIV vaccine, at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the adjusted GMT ratio between FluD-QIVSeq group and FluD-QIVCoAd group for anti-HI antibody titer was <1.5 for the B/Yamagata lineage influenza strain; ANCOVA; GMT Ratio = 1.04, 95% CI 2-sided [0.93 to 1.17]

4. Primary Outcome: Anti-S Protein Antibody Concentrations Expressed as GMCs in FluD-QIVSeq and FluD-QIVCoAd Groups, and Between-group Ratios
Description: Anti-S antibody concentrations were determined by Multiplex Electrochemiluminescence assay and expressed as GMCs in AU/mL.
Time Frame: At 1 month post-mRNA-1273 booster dose administration (Week 4 for both FluD-QIVSeq and FluD-QIVCoAd groups)
Population: mRNA-1273 Per Protocol Set (for Flu D-QIV groups) included all participants who met all eligibility criteria, received all doses as per assignment, for whom administration site of study vaccine was known, who did not receive any other prohibited concomitant intervention, did not meet any of the criteria for elimination during the study through the last blood sample for the group, and with immunogenicity data available for the specified analysis at the specified time point post-mRNA-1273 dose.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 464 | 458
AU/mL | 482604.31 [423492.63 to 549966.87] | 494646.32 [458286.58 to 533890.79]
Statistical Analysis 1: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of mRNA-1273 booster when co-administered with Flu D-QIV vaccine compared to mRNA-1273 booster dose administered alone in terms of anti-S protein GMCs, at 1 month post-mRNA-1273 booster dose administration (at Week 4 for both FluD-QIVSeq and FluD-QIVCoAd groups); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the adjusted GMC ratio between FluD-QIVSeq group and FluD-QIVCoAd group for anti-S antibody concentration was <1.5; ANCOVA; GMC Ratio = 0.98, 95% CI 2-sided [0.84 to 1.13]

5. Secondary Outcome: Percentage of Participants Seroconverted for Anti-HI Antibodies Against the 4 Influenza Strains in Flu D-QIV Vaccine in FluD-QIVSeq and FluD-QIVCoAd Groups, and Between-group Differences
Description: A participant seroconverted for anti-HI antibodies against the 4 influenza strains is defined as a participant having either a pre-vaccination HI titer below (<) 1:10 and a post-vaccination HI titer greater than or equal to (≥) 1:40, or a pre-vaccination HI titer ≥ 1:10 and at least a 4 fold greater post-vaccination HI titer. The 4 influenza strains assessed were A/H1N1 strain, A/H3N2 strain, B/Victoria lineage and B/Yamagata lineage.
Time Frame: At 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 454 | 462
Percentage of participants
  A/H1N1: number analyzed (Participants) | 453 | 461
  A/H1N1 | 73.7 [69.4 to 77.7] | 73.1 [68.8 to 77.1]
  A/H3N2 | 48.7 [44.0 to 53.4] | 50.0 [45.3 to 54.7]
  B/Victoria lineage | 28.9 [24.7 to 33.3] | 28.8 [24.7 to 33.2]
  B/Yamagata lineage | 22.0 [18.3 to 26.1] | 23.6 [19.8 to 27.7]
Statistical Analysis 1: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of Flu D-QIV vaccine when co-administered with mRNA-1273 booster dose compared to Flu D-QIV vaccine administered alone, in terms of percentage of participants seroconverted for anti-HI antibodies against the A/H1N1 influenza strain included in the Flu D-QIV vaccine, at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the difference in percentage of participants seroconverted for anti-HI antibodies against the A/H1N1 influenza strain between FluD-QIVSeq group and FluD-QIVCoAd group was < 10%; ANCOVA; Difference in percentage = 0.6, 95% CI 2-sided [-5.1 to 6.4]
Statistical Analysis 2: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of Flu D-QIV vaccine when co-administered with mRNA-1273 booster dose compared to Flu D-QIV vaccine administered alone, in terms of percentage of participants seroconverted for anti-HI antibodies against the A/H3N2 influenza strain included in the Flu D-QIV vaccine, at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the difference in percentage of participants seroconverted for anti-HI antibodies against the A/H3N2 influenza strain between FluD-QIVSeq group and FluD-QIVCoAd group was < 10%; ANCOVA; Difference in percentage = -1.3, 95% CI 2-sided [-7.8 to 5.2]
Statistical Analysis 3: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of Flu D-QIV vaccine when co-administered with mRNA-1273 booster dose compared to Flu D-QIV vaccine administered alone, in terms of percentage of participants seroconverted for anti-HI antibodies against the B/Victoria lineage influenza strain included in the Flu D-QIV vaccine, at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the difference in percentage of participants seroconverted for anti-HI antibodies against the B/Victoria lineage influenza strain between FluD-QIVSeq group and FluD-QIVCoAd group was < 10%; ANCOVA; Difference in percentage = 0.1, 95% CI 2-sided [-5.8 to 5.9]
Statistical Analysis 4: Comparison: FluD-QIVSeq Group vs FluD-QIVCoAd Group; To demonstrate the non-inferiority of humoral immunogenicity of 1 dose of Flu D-QIV vaccine when co-administered with mRNA-1273 booster dose compared to Flu D-QIV vaccine administered alone, in terms of percentage of participants seroconverted for anti-HI antibodies against the B/Yamagata influenza strain included in the Flu D-QIV vaccine, at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group); Test type: Non-Inferiority — The non-inferiority was to be concluded if the UL of the 95% CI of the difference in percentage of participants seroconverted for anti-HI antibodies against the B/Yamagata influenza strain between FluD-QIVSeq group and FluD-QIVCoAd group was < 10%; ANCOVA; Difference in percentage = -1.6, 95% CI 2-sided [-7.0 to 3.9]

6. Secondary Outcome: Percentage of Participants Seropositive for Anti-gE Antibodies in HZ/suSeq and HZ/suCoAd Groups
Description: A participant seropositive for anti-gE antibodies is defined as a participant whose anti-gE antibody concentration was greater than or equal to the assay cut-off value (97 mIU/mL).
Time Frame: At pre-vaccination (Week 2 for HZ/suSeq group and Day 1 for HZ/suCoAd group) and at 1 month post-dose 2 of HZ/su vaccine administration (Week 14 for HZ/suSeq group and Week 12 for HZ/suCoAd group)
Population: HZ/su Per Protocol Set included all participants who met all eligibility criteria, received all doses as per assignment, for whom administration site of study vaccine was known, who did not receive any other prohibited concomitant intervention, did not meet any of the criteria for elimination up to blood sample collection post-HZ/su Dose 2, and with immunogenicity data available for the specified analysis at the specified time points pre-vaccination and post-HZ/su Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 228 | 230
Percentage of participants
  Pre-vaccination | 96.9 [93.8 to 98.8] | 98.3 [95.6 to 99.5]
  1 month post-HZ/su Dose 2 | 100 [98.4 to 100] | 100 [98.4 to 100]

7. Secondary Outcome: Anti-gE Antibody Concentrations Expressed as GMCs in HZ/suSeq and HZ/suCoAd Groups
Description: Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in mIU/mL.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 228 | 230
mIU/mL
  Pre-vaccination | 1243.79 [1060.96 to 1458.12] | 1361.01 [1195.56 to 1549.36]
  1 month post-HZ/su Dose 2 | 47434.82 [43306.87 to 51956.24] | 47599.82 [43960.57 to 51540.33]

8. Secondary Outcome: Percentage of Participants With a Vaccine Response for Anti-gE in HZ/suSeq and HZ/suCoAd Groups
Description: A participant with vaccine response for anti-gE is defined as a participant with:
  * At least a 4-fold greater post-dose anti-gE antibodies concentration as compared to the pre-vaccination anti-gE antibodies concentration, for participants who were seropositive at pre-vaccination, or,
  * At least a 4-fold greater post-dose anti-gE antibodies concentration as compared to the anti-gE antibodies cut-off value for seropositivity, for participants who were seronegative at pre-vaccination.
Time Frame: At 1 month post-dose 2 of HZ/su vaccine administration (Week 14 for HZ/suSeq group and Week 12 for HZ/suCoAd group)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 228 | 230
Percentage of participants | 96.9 [93.8 to 98.8] | 97.4 [94.4 to 99.0]

9. Secondary Outcome: Mean Geometric Increase (MGI) for Anti-gE in HZ/suSeq and HZ/suCoAd Groups
Description: MGI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-gE antibody concentration to the pre-vaccination anti-gE antibody concentration.
Time Frame: At 1 month post-dose 2 of HZ/su vaccine administration (Week 14 for HZ/suSeq group and Week 12 for HZ/suCoAd group) compared to pre-vaccination (Week 2 for HZ/suSeq group and Day 1 for HZ/suCoAd group)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 228 | 230
Ratio | 38.14 [32.02 to 45.42] | 34.97 [30.37 to 40.27]

10. Secondary Outcome: Anti-S Protein Antibody Concentrations Expressed as GMCs in HZ/suSeq and HZ/suCoAd Groups
Description: as for outcome 4
Time Frame: At pre-vaccination (Day 1) and at 1 month post-mRNA-1273 booster dose administration (Week 4 for both HZ/suSeq and HZ/suCoAd groups)
Population: mRNA-1273 Per Protocol Set (for HZ/su groups) included all participants who met all eligibility criteria, received all doses as per assignment, for whom administration site of study vaccine was known, who did not receive any other prohibited concomitant intervention, did not meet any of the criteria for elimination up to blood sample collection post-mRNA-1273 dose, and with immunogenicity data available for the specified analysis at the specified time points pre- and post-mRNA-1273 dose.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 247 | 247
AU/mL
  Pre-vaccination | 33138.45 [28222.94 to 38910.09] | 34223.23 [29039.32 to 40332.54]
  1 month post-mRNA-1273 booster dose | 618638.92 [526014.86 to 727572.81] | 567728.74 [513530.08 to 627647.61]

11. Secondary Outcome: Anti-S Protein Antibody Concentrations Expressed as GMCs in FluD-QIVSeq and FluD-QIVCoAd Groups
Description: as for outcome 4
Time Frame: At pre-vaccination (Day 1) and at 1 month post-mRNA-1273 booster dose administration (Week 4 for both FluD-QIVSeq and FluD-QIVCoAd groups)
Population: mRNA-1273 Per Protocol Set(for Flu D-QIV groups) included all participants who met all eligibility criteria, received all doses as per assignment, for whom administration site of vaccine was known, who did not receive any other prohibited concomitant intervention, did not meet any of the criteria for elimination during the study through the last blood sample for the group, and with immunogenicity data available for the specified analysis at the specified time points pre- and post-mRNA-1273 dose.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 464 | 458
AU/mL
  Pre-vaccination | 32654.66 [28833.08 to 36982.76] | 33635.52 [29510.93 to 38336.58]
  1 month post-mRNA-1273 booster dose | 482604.31 [423492.63 to 549966.87] | 494646.32 [458286.58 to 533890.79]

12. Secondary Outcome: Mean Geometric Increase (MGI) for Anti-S Protein in HZ/suSeq and HZ/suCoAd Groups
Description: MGI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-S protein antibody concentration to the pre-vaccination anti-S protein antibody concentration.
Time Frame: At 1 month post-mRNA-1273 booster dose administration (Week 4 for both HZ/suSeq and HZ/suCoAd groups) compared to pre-vaccination (Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 247 | 247
Ratio | 18.67 [15.22 to 22.90] | 16.59 [13.73 to 20.04]

13. Secondary Outcome: Mean Geometric Increase (MGI) for Anti-S Protein in FluD-QIVSeq and FluD-QIVCoAd Groups
Description: as for outcome 12
Time Frame: At 1 month post-mRNA-1273 booster dose administration (Week 4 for both FluD-QIVSeq and FluD-QIVCoAd groups) compared to pre-vaccination (Day 1)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 464 | 458
Ratio | 14.78 [12.55 to 17.41] | 14.71 [12.87 to 16.81]

14. Secondary Outcome: Anti-HI Antibody Titers Expressed as GMTs Against the 4 Influenza Strains in Flu D-QIV Vaccine in FluD-QIVSeq and FluD-QIVCoAd Groups
Description: as for outcome 3
Time Frame: At pre-vaccination (Week 2 for FluD-QIVSeq group and Day 1 for FluD-QIVCoAd group) and at 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group)
Population: Flu D-QIV Per Protocol Set included all participants who met all eligibility criteria, received all doses as per assignment, for whom administration site of study vaccine was known, who did not receive any other prohibited concomitant intervention, did not meet any of the criteria for elimination during the study through the last blood sample for the group, and with immunogenicity data available for the specified analysis at the specified time points pre- and post-Flu D-QIV dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 454 | 462
Titers
  A/H1N1, at Pre-vaccination | 65.18 [57.38 to 74.04] | 61.86 [54.18 to 70.64]
  A/H1N1, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 453 | 461
  A/H1N1, at 1 month post-Flu D-QIV dose | 598.62 [535.51 to 669.17] | 577.77 [517.80 to 644.68]
  A/H3N2, at Pre-vaccination | 70.93 [62.14 to 80.97] | 66.30 [58.08 to 75.68]
  A/H3N2, at 1 month post-Flu D-QIV dose | 268.32 [242.17 to 297.30] | 280.26 [252.47 to 311.11]
  B/Victoria lineage, at Pre-vaccination | 17.92 [16.11 to 19.93] | 17.48 [15.78 to 19.37]
  B/Victoria lineage, at 1 month post-Flu D-QIV dose | 48.00 [43.19 to 53.34] | 47.21 [42.47 to 52.49]
  B/Yamagata lineage, at Pre-vaccination | 23.42 [20.92 to 26.23] | 20.49 [18.38 to 22.85]
  B/Yamagata lineage, at 1 month post-Flu D-QIV dose | 55.30 [49.64 to 61.61] | 48.74 [43.83 to 54.21]

15. Secondary Outcome: Percentage of Participants Seroprotected for Anti-HI Antibodies Against the 4 Influenza Strains in FluD-QIV Vaccine in FluD-QIVSeq and FluD-QIVCoAd Groups, Overall and by Age Category
Description: A participant seroprotected for anti-HI antibodies against the 4 influenza strains included in the FluD-QIV vaccine is defined as a participant with a serum HI titer ≥ 1:40. The 4 influenza strains assessed were A/H1N1 strain, A/H3N2 strain, B/Victoria lineage and B/Yamagata lineage. The age categories assessed were 18-64 and ≥ 65 years of age (YOA).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 454 | 462
Percentage of participants
  A/H1N1, overall, at Pre-vaccination | 71.1 [66.7 to 75.3] | 69.3 [64.8 to 73.4]
  A/H1N1, overall, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 453 | 461
  A/H1N1, overall, at 1 month post-Flu D-QIV dose | 98.9 [97.4 to 99.6] | 98.5 [96.9 to 99.4]
  A/H3N2, overall, at Pre-vaccination | 71.1 [66.7 to 75.3] | 69.0 [64.6 to 73.2]
  A/H3N2, overall, at 1 month post-Flu D-QIV dose | 96.9 [94.9 to 98.3] | 95.7 [93.4 to 97.3]
  B/Victoria lineage, overall, at Pre-vaccination | 30.8 [26.6 to 35.3] | 30.1 [25.9 to 34.5]
  B/Victoria lineage, overall, at 1 month post-Flu D-QIV dose | 63.2 [58.6 to 67.7] | 64.7 [60.2 to 69.1]
  B/Yamagata lineage, overall, at Pre-vaccination | 39.9 [35.3 to 44.5] | 36.1 [31.8 to 40.7]
  B/Yamagata lineage, overall, at 1 month post-Flu D-QIV dose | 68.3 [63.8 to 72.5] | 65.6 [61.1 to 69.9]
  A/H1N1, 18-64 YOA category, at Pre-vaccination: number analyzed (Participants) | 358 | 366
  A/H1N1, 18-64 YOA category, at Pre-vaccination | 73.2 [68.3 to 77.7] | 71.6 [66.7 to 76.2]
  A/H1N1, 18-64 YOA category, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 358 | 365
  A/H1N1, 18-64 YOA category, at 1 month post-Flu D-QIV dose | 99.7 [98.5 to 100] | 99.5 [98.0 to 99.9]
  A/H3N2, 18-64 YOA category, at Pre-vaccination: number analyzed (Participants) | 358 | 366
  A/H3N2, 18-64 YOA category, at Pre-vaccination | 72.6 [67.7 to 77.2] | 70.5 [65.5 to 75.1]
  A/H3N2, 18-64 YOA category, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 358 | 366
  A/H3N2, 18-64 YOA category, at 1 month post-Flu D-QIV dose | 98.3 [96.4 to 99.4] | 96.4 [94.0 to 98.1]
  B/Victoria lineage, 18-64 YOA category, at Pre-vaccination: number analyzed (Participants) | 358 | 366
  B/Victoria lineage, 18-64 YOA category, at Pre-vaccination | 29.3 [24.7 to 34.3] | 31.4 [26.7 to 36.4]
  B/Victoria lineage, 18-64 YOA category, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 358 | 366
  B/Victoria lineage, 18-64 YOA category, at 1 month post-Flu D-QIV dose | 64.2 [59.0 to 69.2] | 66.9 [61.9 to 71.7]
  B/Yamagata lineage, 18-64 YOA category, at Pre-vaccination: number analyzed (Participants) | 358 | 366
  B/Yamagata lineage, 18-64 YOA category, at Pre-vaccination | 44.7 [39.5 to 50.0] | 38.5 [33.5 to 43.7]
  B/Yamagata lineage, 18-64 YOA category, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 358 | 366
  B/Yamagata lineage, 18-64 YOA category, at 1 month post-Flu D-QIV dose | 75.1 [70.3 to 79.5] | 69.9 [65.0 to 74.6]
  A/H1N1, ≥65 YOA category, at Pre-vaccination: number analyzed (Participants) | 96 | 96
  A/H1N1, ≥65 YOA category, at Pre-vaccination | 63.5 [53.1 to 73.1] | 60.4 [49.9 to 70.3]
  A/H1N1, ≥65 YOA category, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 95 | 96
  A/H1N1, ≥65 YOA category, at 1 month post-Flu D-QIV dose | 95.8 [89.6 to 98.8] | 94.8 [88.3 to 98.3]
  A/H3N2, ≥65 YOA category, at Pre-vaccination: number analyzed (Participants) | 96 | 96
  A/H3N2, ≥65 YOA category, at Pre-vaccination | 65.6 [55.2 to 75.0] | 63.5 [53.1 to 73.1]
  A/H3N2, ≥65 YOA category, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 96 | 96
  A/H3N2, ≥65 YOA category, at 1 month post-Flu D-QIV dose | 91.7 [84.2 to 96.3] | 92.7 [85.6 to 97.0]
  B/Victoria lineage, ≥65 YOA category, at Pre-vaccination: number analyzed (Participants) | 96 | 96
  B/Victoria lineage, ≥65 YOA category, at Pre-vaccination | 36.5 [26.9 to 46.9] | 25.0 [16.7 to 34.9]
  B/Victoria lineage, ≥65 YOA category, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 96 | 96
  B/Victoria lineage, ≥65 YOA category, at 1 month post-Flu D-QIV dose | 59.4 [48.9 to 69.3] | 56.3 [45.7 to 66.4]
  B/Yamagata lineage, ≥65 YOA category, at Pre-vaccination: number analyzed (Participants) | 96 | 96
  B/Yamagata lineage, ≥65 YOA category, at Pre-vaccination | 21.9 [14.1 to 31.5] | 27.1 [18.5 to 37.1]
  B/Yamagata lineage, ≥65 YOA category, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 96 | 96
  B/Yamagata lineage, ≥65 YOA category, at 1 month post-Flu D-QIV dose | 42.7 [32.7 to 53.2] | 49.0 [38.6 to 59.4]

16. Secondary Outcome: Percentage of Participants Seropositive for Anti-HI Antibodies Against the 4 Influenza Strains in FluD-QIV Vaccine in FluD-QIVSeq and FluD-QIVCoAd Groups
Description: A participant seropositive for anti-HI antibodies against the 4 influenza strains included in the FluD-QIV vaccine is defined as a participant with a serum HI titer ≥ 1:10. The 4 influenza strains assessed were A/H1N1 strain, A/H3N2 strain, B/Victoria lineage and B/Yamagata lineage.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 454 | 462
Percentage of participants
  A/H1N1, at Pre-vaccination | 91.6 [88.7 to 94.0] | 89.8 [86.7 to 92.4]
  A/H1N1, at 1 month post-Flu D-QIV dose: number analyzed (Participants) | 453 | 461
  A/H1N1, at 1 month post-Flu D-QIV dose | 99.8 [98.8 to 100] | 99.8 [98.8 to 100]
  A/H3N2, at Pre-vaccination | 94.5 [92.0 to 96.4] | 92.6 [89.9 to 94.8]
  A/H3N2, at 1 month post-Flu D-QIV dose | 99.8 [98.8 to 100] | 99.4 [98.1 to 99.9]
  B/Victoria lineage, at Pre-vaccination | 70.7 [66.3 to 74.9] | 72.1 [67.7 to 76.1]
  B/Victoria lineage, at 1 month post-Flu D-QIV dose | 94.9 [92.5 to 96.8] | 95.2 [92.9 to 97.0]
  B/Yamagata lineage, at Pre-vaccination | 78.4 [74.3 to 82.1] | 74.7 [70.5 to 78.6]
  B/Yamagata lineage, at 1 month post-Flu D-QIV dose | 96.7 [94.6 to 98.1] | 95.0 [92.6 to 96.8]

17. Secondary Outcome: Mean Geometric Increase (MGI) for Anti-HI Against the 4 Influenza Strains in FluD-QIV Vaccine in FluD-QIVSeq and FluD-QIVCoAd Groups
Description: MGI is defined as the geometric mean of the within participant ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer. The 4 influenza strains assessed were A/H1N1 strain, A/H3N2 strain, B/Victoria lineage and B/Yamagata lineage.
Time Frame: At 1 month post-Flu D-QIV vaccine dose administration (Week 6 for FluD-QIVSeq group and Week 4 for FluD-QIVCoAd group) compared to pre-vaccination (Week 2 for FluD-QIVSeq group and Day 1 for FluD-QIVCoAd group)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 454 | 462
Ratio
  A/H1N1: number analyzed (Participants) | 453 | 461
  A/H1N1 | 9.20 [8.02 to 10.56] | 9.38 [8.13 to 10.82]
  A/H3N2 | 3.78 [3.38 to 4.23] | 4.23 [3.75 to 4.76]
  B/Victoria lineage | 2.68 [2.42 to 2.96] | 2.70 [2.44 to 2.99]
  B/Yamagata lineage | 2.36 [2.16 to 2.58] | 2.38 [2.18 to 2.60]

18. Secondary Outcome: Percentage of Participants Seroconverted for Anti-HI Antibodies Against the 4 Influenza Strains in FluD-QIV Vaccine in FluD-QIVSeq and FluD-QIVCoAd Groups, Overall and by Age Category
Description: A participant seroconverted for anti-HI antibodies against the 4 influenza strains is defined as a participant having either a pre-vaccination HI titer < 1:10 and a post-vaccination HI titer ≥ 1:40, or a pre-vaccination HI titer ≥ 1:10 and at least a 4 fold greater post-vaccination HI titer.
  The 4 influenza strains assessed were A/H1N1 strain, A/H3N2 strain, B/Victoria lineage and B/Yamagata lineage. The age categories assessed were 18-64 and ≥65 years of age (YOA).
Time Frame: as for outcome 17
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 454 | 462
Percentage of participants
  A/H1N1, overall: number analyzed (Participants) | 453 | 461
  A/H1N1, overall | 73.7 [69.4 to 77.7] | 73.1 [68.8 to 77.1]
  A/H3N2, overall | 48.7 [44.0 to 53.4] | 50.0 [45.3 to 54.7]
  B/Victoria lineage, overall | 28.9 [24.7 to 33.3] | 28.8 [24.7 to 33.2]
  B/Yamagata lineage, overall | 22.0 [18.3 to 26.1] | 23.6 [19.8 to 27.7]
  A/H1N1, 18-64 YOA category: number analyzed (Participants) | 358 | 365
  A/H1N1, 18-64 YOA category | 73.7 [68.9 to 78.2] | 75.3 [70.6 to 79.7]
  A/H3N2, 18-64 YOA category: number analyzed (Participants) | 358 | 366
  A/H3N2, 18-64 YOA category | 49.7 [44.4 to 55.0] | 50.8 [45.6 to 56.1]
  B/Victoria lineage, 18-64 YOA category: number analyzed (Participants) | 358 | 366
  B/Victoria lineage, 18-64 YOA category | 31.3 [26.5 to 36.4] | 29.5 [24.9 to 34.5]
  B/Yamagata lineage, 18-64 YOA category: number analyzed (Participants) | 358 | 366
  B/Yamagata lineage, 18-64 YOA category | 23.2 [18.9 to 27.9] | 24.6 [20.3 to 29.3]
  A/H1N1, ≥65 YOA category: number analyzed (Participants) | 95 | 96
  A/H1N1, ≥65 YOA category | 73.7 [63.6 to 82.2] | 64.6 [54.2 to 74.1]
  A/H3N2, ≥65 YOA category: number analyzed (Participants) | 96 | 96
  A/H3N2, ≥65 YOA category | 44.8 [34.6 to 55.3] | 46.9 [36.6 to 57.3]
  B/Victoria lineage, ≥65 YOA category: number analyzed (Participants) | 96 | 96
  B/Victoria lineage, ≥65 YOA category | 19.8 [12.4 to 29.2] | 26.0 [17.6 to 36.0]
  B/Yamagata lineage, ≥65 YOA category: number analyzed (Participants) | 96 | 96
  B/Yamagata lineage, ≥65 YOA category | 17.7 [10.7 to 26.8] | 19.8 [12.4 to 29.2]

19. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Solicited Local Adverse Events (AEs)
Description: The assessed solicited local AEs included axillary (underarm) swelling or tenderness, pain, pruritus, redness and swelling. Axillary swelling or tenderness was solicited for all participants and not restricted to mRNA-1273 recipients as was originally planned per protocol. Pruritus was solicited for all participants and not restricted to HZ/su recipients as was originally planned per protocol.
Time Frame: Within 7 days after each vaccine dose and across doses (vaccines administered at Day 1, Week 2 and Week 10 for HZ/suSeq group and at Day 1 and Week 8 for HZ/suCoAd group)
Population: The HZ/su and mRNA-1273 Exposed set (for solicited safety analysis) included all participants in the HZ/su and mRNA-1273 booster cohort (HZ/suSeq and HZ/suCoAd groups) with at least 1 vaccine administration documented and with the electronic diary completed post-each vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants
  Axillary (underarm) Swelling or Tenderness, Across doses | 15.1 [11.0 to 19.9] | 15.4 [11.3 to 20.2]
  Pain, Across doses | 81.6 [76.5 to 86.0] | 80.9 [75.7 to 85.4]
  Pruritus, Across doses | 25.0 [20.0 to 30.6] | 22.1 [17.3 to 27.6]
  Redness, Across doses | 17.6 [13.3 to 22.7] | 13.5 [9.6 to 18.2]
  Swelling, Across doses | 8.8 [5.7 to 12.8] | 9.7 [6.5 to 13.9]
  Axillary Swelling or Tenderness, post-mRNA-1273 booster dose | 7.0 [4.3 to 10.7] | 7.1 [4.3 to 10.9]
  Pain, post-mRNA-1273 booster dose | 61.8 [55.7 to 67.6] | 63.7 [57.6 to 69.4]
  Pruritus, post-mRNA-1273 booster dose | 10.7 [7.3 to 15.0] | 10.9 [7.4 to 15.2]
  Redness, post-mRNA-1273 booster dose | 4.0 [2.0 to 7.1] | 3.7 [1.8 to 6.8]
  Swelling, post-mRNA-1273 booster dose | 3.7 [1.8 to 6.7] | 3.4 [1.6 to 6.3]
  Axillary Swelling or Tenderness, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 267
  Axillary Swelling or Tenderness, post-HZ/su Dose 1 | 6.5 [3.8 to 10.2] | 6.0 [3.5 to 9.5]
  Pain, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 267
  Pain, post-HZ/su Dose 1 | 64.1 [58.0 to 69.9] | 70.8 [64.9 to 76.2]
  Pruritus, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 267
  Pruritus, post-HZ/su Dose 1 | 10.7 [7.2 to 15.1] | 9.0 [5.8 to 13.1]
  Redness, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 267
  Redness, post-HZ/su Dose 1 | 6.5 [3.8 to 10.2] | 5.2 [2.9 to 8.6]
  Swelling, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 267
  Swelling, post-HZ/su Dose 1 | 2.7 [1.1 to 5.4] | 4.1 [2.1 to 7.3]
  Axillary Swelling or Tenderness, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Axillary Swelling or Tenderness, post-HZ/su Dose 2 | 5.8 [3.3 to 9.4] | 5.8 [3.3 to 9.4]
  Pain, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Pain, post-HZ/su Dose 2 | 58.5 [52.3 to 64.6] | 59.1 [52.9 to 65.2]
  Pruritus, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Pruritus, post-HZ/su Dose 2 | 12.8 [9.0 to 17.5] | 13.2 [9.3 to 18.0]
  Redness, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Redness, post-HZ/su Dose 2 | 11.2 [7.7 to 15.7] | 9.3 [6.1 to 13.6]
  Swelling, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Swelling, post-HZ/su Dose 2 | 5.0 [2.7 to 8.5] | 5.4 [3.0 to 9.0]

20. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Reporting Solicited Local Adverse Events (AEs)
Description: as for outcome 19
Time Frame: Within 7 days after each vaccine dose and across doses (vaccines administered at Day 1 and Week 2 for FluD-QIVSeq group and at Day 1 for FluD-QIVCoAd group)
Population: The Flu D-QIV and mRNA-1273 Exposed set (for solicited safety analysis) included all participants in the Flu D-QIV and mRNA-1273 booster cohort (FluD-QIVSeq and FluD-QIVCoAd groups) with at least 1 vaccine administration documented and with the electronic diary completed post-each vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 496 | 497
Percentage of participants
  Axillary (underarm) Swelling or Tenderness, Across doses | 20.0 [16.5 to 23.8] | 14.3 [11.3 to 17.7]
  Pain, Across doses | 77.8 [73.9 to 81.4] | 74.6 [70.6 to 78.4]
  Pruritus, Across doses | 13.9 [11.0 to 17.3] | 13.9 [11.0 to 17.2]
  Redness, Across doses | 7.9 [5.7 to 10.6] | 5.4 [3.6 to 7.8]
  Swelling, Across doses | 6.5 [4.5 to 9.0] | 6.0 [4.1 to 8.5]
  Axillary Swelling or Tenderness, post-mRNA-1273 booster dose | 16.3 [13.2 to 19.9] | 12.5 [9.7 to 15.7]
  Pain, post-mRNA-1273 booster dose | 75.8 [71.8 to 79.5] | 71.8 [67.7 to 75.7]
  Pruritus, post-mRNA-1273 booster dose | 12.1 [9.4 to 15.3] | 11.9 [9.2 to 15.0]
  Redness, post-mRNA-1273 booster dose | 7.1 [5.0 to 9.7] | 4.8 [3.1 to 7.1]
  Swelling, post-mRNA-1273 booster dose | 6.0 [4.1 to 8.5] | 5.6 [3.8 to 8.0]
  Axillary Swelling or Tenderness, post-Flu D-QIV dose: number analyzed (Participants) | 490 | 497
  Axillary Swelling or Tenderness, post-Flu D-QIV dose | 5.7 [3.8 to 8.2] | 6.6 [4.6 to 9.2]
  Pain, post-Flu D-QIV dose: number analyzed (Participants) | 490 | 497
  Pain, post-Flu D-QIV dose | 30.6 [26.6 to 34.9] | 48.1 [43.6 to 52.6]
  Pruritus, post-Flu D-QIV dose: number analyzed (Participants) | 490 | 497
  Pruritus, post-Flu D-QIV dose | 4.5 [2.8 to 6.7] | 3.8 [2.3 to 5.9]
  Redness, post-Flu D-QIV dose: number analyzed (Participants) | 490 | 497
  Redness, post-Flu D-QIV dose | 1.8 [0.8 to 3.5] | 0.8 [0.2 to 2.0]
  Swelling, post-Flu D-QIV dose: number analyzed (Participants) | 490 | 497
  Swelling, post-Flu D-QIV dose | 1.0 [0.3 to 2.4] | 1.2 [0.4 to 2.6]

21. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Solicited Systemic Adverse Events (AEs)
Description: The assessed solicited systemic AEs included abdominal pain, arthralgia, chills, diarrhea, fatigue, fever, gastrointestinal symptoms, headache, myalgia, nausea and vomiting. Fever is defined as temperature ≥ 38.0 degrees Celsius (°C)/100.4 degrees Fahrenheit (°F) by any route. The preferred location for measuring temperature was the oral route.
Time Frame: as for outcome 19
Population: The HZ/su and mRNA-1273 Exposed set (for solicited safety analysis) included all participants in the HZ/su and mRNA-1273 booster cohort (HZ/suSeq and HZ/suCoAd groups) with at least 1 vaccine administration documented and with the electronic diary completed post-each vaccination. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants
  Abdominal Pain, Across doses | 11.0 [7.6 to 15.4] | 12.4 [8.7 to 16.9]
  Arthralgia, Across doses | 37.5 [31.7 to 43.5] | 40.8 [34.9 to 47.0]
  Chills, Across doses | 39.0 [33.1 to 45.0] | 40.1 [34.1 to 46.2]
  Diarrhea, Across doses | 20.6 [15.9 to 25.9] | 19.5 [14.9 to 24.7]
  Fatigue, Across doses | 56.3 [50.1 to 62.2] | 60.3 [54.2 to 66.2]
  Fever, Across doses | 10.7 [7.3 to 15.0] | 13.1 [9.3 to 17.8]
  Gastrointestinal Symptoms, Across doses | 34.9 [29.3 to 40.9] | 34.1 [28.4 to 40.1]
  Headache, Across doses | 46.3 [40.3 to 52.4] | 51.3 [45.1 to 57.4]
  Myalgia, Across doses | 65.4 [59.5 to 71.1] | 72.7 [66.9 to 77.9]
  Nausea, Across doses | 18.8 [14.3 to 23.9] | 16.9 [12.6 to 21.9]
  Vomiting, Across doses | 2.9 [1.3 to 5.7] | 3.7 [1.8 to 6.8]
  Abdominal Pain, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Abdominal Pain, post-HZ/su Dose 1 | 2.7 [1.1 to 5.4] |
  Arthralgia, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Arthralgia, post-HZ/su Dose 1 | 19.1 [14.5 to 24.4] |
  Chills, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Chills, post-HZ/su Dose 1 | 14.9 [10.8 to 19.8] |
  Diarrhea, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Diarrhea, post-HZ/su Dose 1 | 6.9 [4.1 to 10.6] |
  Fatigue, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Fatigue, post-HZ/su Dose 1 | 32.1 [26.5 to 38.1] |
  Fever, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Fever, post-HZ/su Dose 1 | 3.8 [1.8 to 6.9] |
  Gastrointestinal Symptoms, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Gastrointestinal Symptoms, post-HZ/su Dose 1 | 12.6 [8.8 to 17.2] |
  Headache, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Headache, post-HZ/su Dose 1 | 21.4 [16.6 to 26.8] |
  Myalgia, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Myalgia, post-HZ/su Dose 1 | 37.8 [31.9 to 44.0] |
  Nausea, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Nausea, post-HZ/su Dose 1 | 6.5 [3.8 to 10.2] |
  Vomiting, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Vomiting, post-HZ/su Dose 1 | 0.0 [0.0 to 1.4] |
  Abdominal Pain, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Abdominal Pain, post-HZ/su Dose 2 | 3.5 [1.6 to 6.5] | 6.6 [3.9 to 10.4]
  Arthralgia, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Arthralgia, post-HZ/su Dose 2 | 20.9 [16.1 to 26.4] | 23.3 [18.3 to 29.0]
  Chills, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Chills, post-HZ/su Dose 2 | 21.7 [16.8 to 27.2] | 23.3 [18.3 to 29.0]
  Diarrhea, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Diarrhea, post-HZ/su Dose 2 | 8.5 [5.4 to 12.6] | 10.5 [7.0 to 14.9]
  Fatigue, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Fatigue, post-HZ/su Dose 2 | 32.9 [27.2 to 39.0] | 37.7 [31.8 to 44.0]
  Fever, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Fever, post-HZ/su Dose 2 | 3.9 [1.9 to 7.0] | 4.3 [2.2 to 7.5]
  Gastrointestinal Symptoms, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Gastrointestinal Symptoms, post-HZ/su Dose 2 | 17.1 [12.7 to 22.2] | 19.5 [14.8 to 24.8]
  Headache, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Headache, post-HZ/su Dose 2 | 28.3 [22.9 to 34.2] | 31.9 [26.3 to 38.0]
  Myalgia, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Myalgia, post-HZ/su Dose 2 | 41.9 [35.8 to 48.1] | 43.6 [37.4 to 49.9]
  Nausea, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Nausea, post-HZ/su Dose 2 | 8.1 [5.1 to 12.2] | 9.7 [6.4 to 14.0]
  Vomiting, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Vomiting, post-HZ/su Dose 2 | 1.6 [0.4 to 3.9] | 1.2 [0.2 to 3.4]
  Abdominal Pain, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Abdominal Pain, post-mRNA-1273 booster dose | 5.9 [3.4 to 9.4] |
  Arthralgia, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Arthralgia, post-mRNA-1273 booster dose | 22.4 [17.6 to 27.9] |
  Chills, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Chills, post-mRNA-1273 booster dose | 19.5 [14.9 to 24.7] |
  Diarrhea, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Diarrhea, post-mRNA-1273 booster dose | 12.1 [8.5 to 16.6] |
  Fatigue, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Fatigue, post-mRNA-1273 booster dose | 36.4 [30.7 to 42.4] |
  Fever, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Fever, post-mRNA-1273 booster dose | 5.1 [2.8 to 8.5] |
  Gastrointestinal Symptoms, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Gastrointestinal Symptoms, post-mRNA-1273 booster dose | 21.0 [16.3 to 26.3] |
  Headache, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Headache, post-mRNA-1273 booster dose | 29.4 [24.1 to 35.2] |
  Myalgia, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Myalgia, post-mRNA-1273 booster dose | 45.6 [39.6 to 51.7] |
  Nausea, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Nausea, post-mRNA-1273 booster dose | 9.9 [6.6 to 14.1] |
  Vomiting, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Vomiting, post-mRNA-1273 booster dose | 1.5 [0.4 to 3.7] |
  Abdominal Pain, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Abdominal Pain, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 7.9 [4.9 to 11.8]
  Arthralgia, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Arthralgia, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 30.3 [24.9 to 36.2]
  Chills, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Chills, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 31.5 [25.9 to 37.4]
  Diarrhea, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Diarrhea, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 13.5 [9.6 to 18.2]
  Fatigue, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Fatigue, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 51.7 [45.5 to 57.8]
  Fever, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Fever, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 10.1 [6.8 to 14.4]
  Gastrointestinal Symptoms, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Gastrointestinal Symptoms, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 24.0 [19.0 to 29.6]
  Headache, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Headache, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 39.0 [33.1 to 45.1]
  Myalgia, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Myalgia, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 64.0 [58.0 to 69.8]
  Nausea, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Nausea, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 10.1 [6.8 to 14.4]
  Vomiting, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Vomiting, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 3.0 [1.3 to 5.8]

22. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Reporting Solicited Systemic Adverse Events (AEs)
Description: The assessed solicited systemic AEs included abdominal pain, arthralgia, chills, diarrhea, fatigue, fever, gastrointestinal symptoms, headache, myalgia, nausea and vomiting. Fever is defined as temperature ≥ 38.0°C/100.4°F by any route. The preferred location for measuring temperature was the oral route.
Time Frame: as for outcome 20
Population: The Flu D-QIV and mRNA-1273 Exposed set (for solicited safety analysis) included all participants in the Flu D-QIV and mRNA-1273 booster cohort (FluD-QIVSeq and FluD-QIVCoAd groups) with at least 1 vaccine administration documented and with the electronic diary completed post-each vaccination. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 496 | 497
Percentage of participants
  Abdominal Pain, Across doses | 10.5 [7.9 to 13.5] | 6.6 [4.6 to 9.2]
  Arthralgia, Across doses | 30.8 [26.8 to 35.1] | 29.8 [25.8 to 34.0]
  Chills, Across doses | 33.1 [28.9 to 37.4] | 29.2 [25.2 to 33.4]
  Diarrhea, Across doses | 24.0 [20.3 to 28.0] | 16.1 [13.0 to 19.6]
  Fatigue, Across doses | 63.7 [59.3 to 67.9] | 57.7 [53.3 to 62.1]
  Fever, Across doses | 6.0 [4.1 to 8.5] | 5.8 [3.9 to 8.3]
  Gastrointestinal Symptoms, Across doses | 39.5 [35.2 to 44.0] | 27.8 [23.9 to 31.9]
  Headache, Across doses | 51.0 [46.5 to 55.5] | 46.7 [42.2 to 51.2]
  Myalgia, Across doses | 64.3 [59.9 to 68.5] | 58.8 [54.3 to 63.1]
  Nausea, Across doses | 21.4 [17.8 to 25.2] | 12.9 [10.1 to 16.1]
  Vomiting, Across doses | 3.2 [1.9 to 5.2] | 1.6 [0.7 to 3.1]
  Abdominal Pain, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Abdominal Pain, post-FluD-QIV dose | 2.9 [1.6 to 4.7] |
  Arthralgia, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Arthralgia, post-FluD-QIV dose | 6.7 [4.7 to 9.3] |
  Chills, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Chills, post-FluD-QIV dose | 6.3 [4.3 to 8.9] |
  Diarrhea, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Diarrhea, post-FluD-QIV dose | 10.6 [8.0 to 13.7] |
  Fatigue, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Fatigue, post-FluD-QIV dose | 19.6 [16.2 to 23.4] |
  Fever, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Fever, post-FluD-QIV dose | 0.8 [0.2 to 2.1] |
  Gastrointestinal Symptoms, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Gastrointestinal Symptoms, post-FluD-QIV dose | 15.9 [12.8 to 19.5] |
  Headache, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Headache, post-FluD-QIV dose | 19.6 [16.2 to 23.4] |
  Myalgia, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Myalgia, post-FluD-QIV dose | 14.5 [11.5 to 17.9] |
  Nausea, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Nausea, post-FluD-QIV dose | 5.7 [3.8 to 8.2] |
  Vomiting, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Vomiting, post-FluD-QIV dose | 1.0 [0.3 to 2.4] |
  Abdominal Pain, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Abdominal Pain, post-mRNA-1273 booster dose | 8.5 [6.2 to 11.3] |
  Arthralgia, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Arthralgia, post-mRNA-1273 booster dose | 28.6 [24.7 to 32.8] |
  Chills, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Chills, post-mRNA-1273 booster dose | 29.6 [25.6 to 33.9] |
  Diarrhea, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Diarrhea, post-mRNA-1273 booster dose | 16.5 [13.4 to 20.1] |
  Fatigue, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Fatigue, post-mRNA-1273 booster dose | 58.5 [54.0 to 62.8] |
  Fever, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Fever, post-mRNA-1273 booster dose | 5.2 [3.5 to 7.6] |
  Gastrointestinal Symptoms, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Gastrointestinal Symptoms, post-mRNA-1273 booster dose | 31.7 [27.6 to 35.9] |
  Headache, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Headache, post-mRNA-1273 booster dose | 46.2 [41.7 to 50.7] |
  Myalgia, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Myalgia, post-mRNA-1273 booster dose | 62.1 [57.7 to 66.4] |
  Nausea, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Nausea, post-mRNA-1273 booster dose | 19.2 [15.8 to 22.9] |
  Vomiting, post-mRNA-1273 booster dose: number analyzed (Participants) | 496 | 0
  Vomiting, post-mRNA-1273 booster dose | 2.2 [1.1 to 3.9] |
  Abdominal Pain, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Abdominal Pain, post-mRNA-1273 booster dose + FluD-QIV dose |  | 6.6 [4.6 to 9.2]
  Arthralgia, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Arthralgia, post-mRNA-1273 booster dose + FluD-QIV dose |  | 29.8 [25.8 to 34.0]
  Chills, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Chills, post-mRNA-1273 booster dose + FluD-QIV dose |  | 29.2 [25.2 to 33.4]
  Diarrhea, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Diarrhea, post-mRNA-1273 booster dose + FluD-QIV dose |  | 16.1 [13.0 to 19.6]
  Fatigue, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Fatigue, post-mRNA-1273 booster dose + FluD-QIV dose |  | 57.7 [53.3 to 62.1]
  Fever, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Fever, post-mRNA-1273 booster dose + FluD-QIV dose |  | 5.8 [3.9 to 8.3]
  Gastrointestinal Symptoms, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Gastrointestinal Symptoms, post-mRNA-1273 booster dose + FluD-QIV dose |  | 27.8 [23.9 to 31.9]
  Headache, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Headache, post-mRNA-1273 booster dose + FluD-QIV dose |  | 46.7 [42.2 to 51.2]
  Myalgia, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Myalgia, post-mRNA-1273 booster dose + FluD-QIV dose |  | 58.8 [54.3 to 63.1]
  Nausea, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Nausea, post-mRNA-1273 booster dose + FluD-QIV dose |  | 12.9 [10.1 to 16.1]
  Vomiting, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 497
  Vomiting, post-mRNA-1273 booster dose + FluD-QIV dose |  | 1.6 [0.7 to 3.1]

23. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as any AE that was either not included in the list of solicited events using a participant diary, or was included in the list of solicited events, but with an onset more than 7 days following administration of a study intervention.
Time Frame: Within 14 days after each vaccine dose and across doses (vaccines administered at Day 1, Week 2 and Week 10 for HZ/suSeq group and at Day 1 and Week 8 for HZ/suCoAd group)
Population: The HZ/su and mRNA-1273 Exposed set (for unsolicited safety analysis) included all participants in the HZ/su and mRNA-1273 booster cohort (HZ/suSeq and HZ/suCoAd groups) with at least 1 vaccine administration documented and with unsolicited AEs data available for the specified duration post-vaccination. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants
  Unsolicited AEs, Across doses | 31.6 [26.1 to 37.5] | 28.8 [23.5 to 34.7]
  Unsolicited AEs, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Unsolicited AEs, post-HZ/su Dose 1 | 14.5 [10.5 to 19.4] |
  Unsolicited AEs, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Unsolicited AEs, post-HZ/su Dose 2 | 10.1 [6.7 to 14.4] | 14.8 [10.7 to 19.7]
  Unsolicited AEs, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Unsolicited AEs, post-mRNA-1273 booster dose | 22.8 [17.9 to 28.2] |
  Unsolicited AEs, post-mRNA-1273 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Unsolicited AEs, post-mRNA-1273 booster dose + HZ/su Dose 1 |  | 20.6 [15.9 to 26.0]

24. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Reporting Unsolicited Adverse Events (AEs)
Description: as for outcome 23
Time Frame: Within 14 days after each vaccine dose and across doses (vaccines administered at Day 1 and Week 2 for FluD-QIVSeq group and at Day 1 for FluD-QIVCoAd group)
Population: The Flu D-QIV and mRNA-1273 Exposed set (for unsolicited safety analysis) included all participants in the Flu D-QIV and mRNA-1273 booster cohort (FluD-QIVSeq and FluD-QIVCoAd groups) with at least 1 vaccine administration documented and with unsolicited AEs data available for the specified duration post-vaccination. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 497 | 498
Percentage of participants
  Unsolicited AEs, Across doses | 35.2 [31.0 to 39.6] | 25.1 [21.3 to 29.2]
  Unsolicited AEs, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Unsolicited AEs, post-FluD-QIV dose | 16.9 [13.7 to 20.6] |
  Unsolicited AEs, post-mRNA-1273 booster dose: number analyzed (Participants) | 497 | 0
  Unsolicited AEs, post-mRNA-1273 booster dose | 26.2 [22.3 to 30.3] |
  Unsolicited AEs, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 498
  Unsolicited AEs, post-mRNA-1273 booster dose + FluD-QIV dose |  | 25.1 [21.3 to 29.2]

25. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Unsolicited Adverse Events (AEs)
Description: as for outcome 23
Time Frame: Within 30 days after each vaccine dose and across vaccine doses (vaccines administered at Day 1, Week 2 and Week 10 for HZ/suSeq group and at Day 1 and Week 8 for HZ/suCoAd group)
Population: The HZ/su and mRNA-1273 Exposed set (for unsolicited safety analysis) included all participants in the HZ/su and mRNA-1273 booster cohort (HZ/suSeq and HZ/suCoAd groups) with at least 1 vaccine administration documented and with unsolicited AEs data available for the specified duration post-vaccination. Here, 'number analyzed' = participants with data available for each specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants
  Unsolicited AEs, Across doses | 41.5 [35.6 to 47.6] | 46.1 [40.0 to 52.2]
  Unsolicited AEs, post-HZ/su Dose 1: number analyzed (Participants) | 262 | 0
  Unsolicited AEs, post-HZ/su Dose 1 | 25.2 [20.1 to 30.9] |
  Unsolicited AEs, post-HZ/su Dose 2: number analyzed (Participants) | 258 | 257
  Unsolicited AEs, post-HZ/su Dose 2 | 15.1 [11.0 to 20.1] | 23.3 [18.3 to 29.0]
  Unsolicited AEs, post-mRNA-1273 booster dose: number analyzed (Participants) | 272 | 0
  Unsolicited AEs, post-mRNA-1273 booster dose | 25.0 [20.0 to 30.6] |
  Unsolicited AEs, post-mRNA-1237 booster dose + HZ/su Dose 1: number analyzed (Participants) | 0 | 267
  Unsolicited AEs, post-mRNA-1237 booster dose + HZ/su Dose 1 |  | 37.1 [31.3 to 43.2]

26. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Reporting Unsolicited Adverse Events (AEs)
Description: as for outcome 23
Time Frame: Within 30 days after each vaccine dose and across vaccine doses (vaccines administered at Day 1 and Week 2 for FluD-QIVSeq group and at Day 1 for FluD-QIVCoAd group)
Population: The Flu D-QIV and mRNA-1273 Exposed set (for unsolicited safety analysis) included all participants in the Flu D-QIV and mRNA-1273 booster cohort (FluD-QIVSeq and FluD-QIVCoAd groups) with at least 1 vaccine administration documented and with unsolicited AEs data available for the specified duration post-vaccination. Here, 'number analyzed' = participants with data available for each specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 497 | 498
Percentage of participants
  Unsolicited AEs, Across doses | 43.1 [38.7 to 47.5] | 36.9 [32.7 to 41.4]
  Unsolicited AEs, post-FluD-QIV dose: number analyzed (Participants) | 490 | 0
  Unsolicited AEs, post-FluD-QIV dose | 27.3 [23.4 to 31.5] |
  Unsolicited AEs, post-mRNA-1273 booster dose: number analyzed (Participants) | 497 | 0
  Unsolicited AEs, post-mRNA-1273 booster dose | 29.6 [25.6 to 33.8] |
  Unsolicited AEs, post-mRNA-1273 booster dose + FluD-QIV dose: number analyzed (Participants) | 0 | 498
  Unsolicited AEs, post-mRNA-1273 booster dose + FluD-QIV dose |  | 36.9 [32.7 to 41.4]

27. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant, was considered or defined as an important medical event, or abnormal pregnancy outcomes.
Time Frame: From first vaccine dose (Day 1) up to 30 days post-last vaccine dose within each group
Population: The HZ/su and mRNA-1273 Exposed set included all participants in the HZ/su and mRNA-1273 booster cohort (HZ/suSeq and HZ/suCoAd groups) with at least 1 vaccine administration documented.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants | 1.5 [0.4 to 3.7] | 1.5 [0.4 to 3.8]

28. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Serious Adverse Events (SAEs)
Description: as for outcome 27
Time Frame: From first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose)
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants | 1.8 [0.6 to 4.2] | 2.2 [0.8 to 4.8]

29. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Reporting Serious Adverse Events (SAEs)
Description: as for outcome 27
Time Frame: From first vaccine dose (Day 1) up to 30 days post-last vaccine dose within each group
Population: The Flu D-QIV and mRNA-1273 Exposed set included all participants in the Flu D-QIV and mRNA-1273 booster cohort (FluD-QIVSeq and FluD-QIVCoAd groups) with at least 1 vaccine administration documented.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 497 | 498
Percentage of participants | 0.2 [0.0 to 1.1] | 0.2 [0.0 to 1.1]

30. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Reporting Serious Adverse Events (SAEs)
Description: as for outcome 27
Time Frame: From first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose)
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 497 | 498
Percentage of participants | 1.4 [0.6 to 2.9] | 0.4 [0.0 to 1.4]

31. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Potential Immune Mediated Diseases (pIMDs)
Description: The assessed pIMDs included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have had an autoimmune etiology.
Time Frame: From first vaccine dose (Day 1) up to 30 days post-last vaccine dose within each group
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants | 0.3 | 0.3

32. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Potential Immune Mediated Diseases (pIMDs)
Description: as for outcome 31
Time Frame: From first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants | 0.3 | 0.3

33. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Adverse Events of Special Interest (AESIs)
Description: AESIs were defined as medical concepts that may have been related to COVID-19 or were of interest in COVID-19 vaccine safety surveillance.
Time Frame: From first vaccine dose (Day 1) up to 30 days post-last vaccine dose within each group
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants | 1.1 | 0.0

34. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Adverse Events of Special Interest (AESIs)
Description: as for outcome 33
Time Frame: From first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants | 1.1 | 0.7

35. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Reporting Adverse Events of Special Interest (AESIs)
Description: as for outcome 33
Time Frame: From first vaccine dose (Day 1) up to 30 days post-last vaccine dose within each group
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 497 | 498
Percentage of participants | 0.0 | 0.0

36. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Reporting Adverse Events of Special Interest (AESIs)
Description: as for outcome 33
Time Frame: From first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose)
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 497 | 498
Percentage of participants | 0.0 | 0.2

37. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Reporting Clinically Suspected HZ Episodes
Description: A suspected HZ episode is defined as a new unilateral rash accompanied by pain broadly defined to include allodynia, pruritus or other sensations without alternative diagnosis.
Time Frame: From first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants | 0.7 | 0.0

38. Secondary Outcome: Percentage of Participants in HZ/suSeq and HZ/suCoAd Groups Meeting Case Definitions of COVID-19
Description: Primary Case Definition: Experienced at least TWO of following systemic symptoms: fever (temperature ≥38ºC), chills, myalgia, headache, sore throat, new olfactory & taste disorder(s), OR at least ONE of following respiratory signs: cough, shortness of breath or difficulty breathing, OR clinical or radiographical evidence of pneumonia; AND must have at least one nasopharyngeal (NP) or nasal swab, or saliva or respiratory sample positive for SARS-CoV-2 by PCR.
  Secondary Case Definition: Following systemic symptoms: fever, or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle aches or body aches, headache, new loss of taste or smell, sore throat, nasal congestion or rhinorrhea, nausea or vomiting, or diarrhea AND a positive NP or nasal swab, or saliva or respiratory sample for SARS-CoV-2 by PCR.
  Tertiary Case Definition: Documented COVID-19 diagnosis made by health care provider and not meeting the above case definitions.
Time Frame: From first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group
Number analyzed (Participants) | 272 | 267
Percentage of participants
  Primary Case Definition | 4.4 | 4.1
  Secondary Case Definition | 2.2 | 2.2
  Tertiary Case Definition | 0.7 | 0.3

39. Secondary Outcome: Percentage of Participants in FluD-QIVSeq and FluD-QIVCoAd Groups Meeting Case Definitions of COVID-19
Description: as for outcome 38
Time Frame: From first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose)
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
Number analyzed (Participants) | 497 | 498
Percentage of participants
  Primary Case Definition | 4.6 | 3.2
  Secondary Case Definition | 1.8 | 2.0
  Tertiary Case Definition | 0.6 | 0.6

ADVERSE EVENTS:
Time Frame: Solicited local and systemic AEs: during the 7-day (Days 1-7) follow-up period after vaccination; Unsolicited AEs: during the 30-day (Days 1-30) follow-up period after vaccination; SAEs: from first vaccine dose (Day 1) up to study end (24 weeks post-last vaccine dose).
Arm/Group | HZ/suSeq Group | HZ/suCoAd Group | FluD-QIVSeq Group | FluD-QIVCoAd Group
All-Cause Mortality (participants affected / at risk) | 0/272 | 0/267 | 0/497 | 0/498
Serious Adverse Events (participants affected / at risk) | 5/272 | 6/267 | 7/497 | 2/498
Other Adverse Events (participants affected / at risk) | 248/272 | 243/267 | 463/497 | 445/498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/suSeq Group (N=272) | HZ/suCoAd Group (N=267) | FluD-QIVSeq Group (N=497) | FluD-QIVCoAd Group (N=498)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendix adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Negative pressure pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HZ/suSeq Group (N=272) | HZ/suCoAd Group (N=267) | FluD-QIVSeq Group (N=497) | FluD-QIVCoAd Group (N=498)
Injection site pain (General disorders) | 222 | 216 | 386 | 371
Fatigue (General disorders) | 157 | 167 | 332 | 302
Chills (General disorders) | 116 | 116 | 179 | 156
Injection site erythema (General disorders) | 49 | 36 | 39 | 27
Pyrexia (General disorders) | 31 | 36 | 32 | 29
Injection site swelling (General disorders) | 25 | 26 | 32 | 30
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 181 | 198 | 330 | 303
Arthralgia (Musculoskeletal and connective tissue disorders) | 115 | 113 | 168 | 161
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 141 | 152 | 284 | 262
Migraine (Nervous system disorders) | 1 | 1 | 0 | 1
Anosmia (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Thoracic outlet syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 68 | 71 | 152 | 125
Nausea (Gastrointestinal disorders) | 62 | 53 | 128 | 93
Abdominal pain (Gastrointestinal disorders) | 39 | 43 | 69 | 47
Vomiting (Gastrointestinal disorders) | 12 | 12 | 32 | 19
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Injection site pruritus (Skin and subcutaneous tissue disorders) | 68 | 59 | 69 | 69
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 42 | 42 | 99 | 72
COVID-19 (Infections and infestations) | 3 | 5 | 6 | 1
Urinary tract infection (Infections and infestations) | 2 | 5 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 1 | 9 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 1 | 1
Administration site pustule (Infections and infestations) | 0 | 1 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 2 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Nasal herpes (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 5 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 1 | 1 | 0
Pseudomonas test positive (Investigations) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Tissue infiltration (General disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 2 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Trunk injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05047770/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT05047770/SAP_001.pdf